CLINICAL TRIAL: NCT05816980
Title: External Beam Radiotherapy for Pelvic Recurrences in Rectal Cancer Patients Previously Treated With Radiotherapy
Brief Title: Re-irradiation for Pelvic Recurrences in Rectal Cancer Patients
Acronym: Re-RAD-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Karen-Lise Garm Spindler, Associate Professor, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFE-1506
Record Dates: First submitted 2016-10-24; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer; Recurrence; Radiation Toxicity
MeSH Terms: conditions — Rectal Neoplasms; Recurrence; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Patients are enrolled according to protocol criteria for hyperfractionated IMRT re-irradiation.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Other): Re-irradiation consisting of hyperfractionated IMRT, 40.8 Gy in 1.2 fractions twice daily 5/7 days weekly, with oral capecitabine 825 mg/m2 BID on radiotherapy treatment days. Re-staging performed 4-6 weeks after the last dose, followed by surgery, when feasible.
  Interventions: Radiation: Hyperfractionated external beam radiation

INTERVENTIONS:
Radiation: Hyperfractionated external beam radiation — 40.8Gy/34 fractions (1.2Gy BID 5/7 days with minimum 6 hours interval) Concurrent capecitabine (825 mg/m2 BID 5/7 days)

SUMMARY:
This study investigates the potential benefit of re-irradiation of patients with locally advanced rectal recurrences, by a prospective phase II clinical, imaging and translational research study.

DETAILED DESCRIPTION:
The overall purpose of this trial is to evaluate the efficacy of re-irradiation of patients with locally advanced rectal cancer (LRRC) recurrences who previously received pelvic irradiation. Patients with potentially resectable LRRC will be treated with hyperfractionated Intensity-Modulated Radiotherapy consisting of 40.8 Gy in 1.2 fractions twice daily with concomitant oral capecitabine followed by surgery, when feasible.

ELIGIBILITY:
Inclusion Criteria:

* Locally recurrent rectal cancer
* Previous pelvic RT for rectal cancer and surgery
* Potentially resectable by MRI and palpation by MDT evaluation
* Absence of non-resectable distant metastases by PET-CT
* Age ≥ 18
* Adequate organ function
* Acceptable bowel and bladder function
* Acceptance for TR sampling

Exclusion Criteria:

* Central small recurrences deemed immediate resectable
* Previous radiotherapy <12 month prior to recurrence
* Non-resectable systemic or regional disease
* Unable to undergo MRI or PET-CT
* Medical comorbidities precluding radical surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Resection rate | At surgery
  Rate of complete pathological resection R0

SECONDARY OUTCOMES:
Physician reported Toxicity | Acute and late toxicity evaluations during and at 6,12 and 36 months post surgery
  Clinical and laboratory AEs (Adverse Events) will be graded according to NCICTCAE (version 4.0).
QoL assessment according to QLQ-CR29 | Pre-treatment and 12 months post surgery
  Assesment of QoL according to EORTC guidelines. The EORTC QLQ-CR29 is a tumor-specific health related QoL questionnaire module for CRC patients. Patients are asked to indicate their symptoms during the past week(s). According to EORTC guidelines, scores can be reported as frequencies of raw scores or scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
QoL assessment according to EORTC QLQ-C30 | Pre-treatment and 12 months post surgery
  Assesment of QoL according to EORTC guidelines. The EORTC QLQ-CR30 is a general health related QoL questionnaire. Patients are asked to indicate their symptoms during the past week(s). According to EORTC guidelines, scores can be reported as frequencies of raw scores or scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
Recurrence rate | Rate of re-recurrence at 6, 12 and 36 months post surgery.
  Rate of re-recurrence
Comparative dose planning study | The VMAT plans generated before treatment start (baseline) is compared to IMPT plans.
  Potential organ at risk sparing when comparing photons vs protons - comparative dose planning

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, MD, Phd, Principal Investigator — Aarhus University Hospital, Depart. Oncology
Locations (2):
- Aarhus University Hospital, Aarhus, Denmark
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
IPDs will not be available to other researchers according to National General data protection regulations. However, data will be published according to guidelines.